CLINICAL TRIAL: NCT03543332
Title: Physical Activity After Cardiac Arrest; Protocol of a Sub-study in the Targeted Hypothermia Versus Targeted Normothermia After Out-of-Hospital Cardiac Arrest Trial (TTM2)
Brief Title: Physical Activity After Cardiac Arrest; a Sub-study in the Target Temperature Management Trial 2
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Halmstad County Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiac Arrest Physical
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Heart Arrest, Out-Of-Hospital; Physical Activity
Keywords: Physical training; Kinesiophobia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac arrest
  Interventions: Diagnostic Test: Measures of physical activity and kinesiophobia
- Myocardial infarction: Myocardial infarction without cardiac arrest
  Interventions: Diagnostic Test: Measures of physical activity and kinesiophobia

INTERVENTIONS:
Diagnostic Test: Measures of physical activity and kinesiophobia — Groups will be compared regarding kinesiophobia with TSK heart.

SUMMARY:
The Target Temperature Management trial 2 (TTM2) is an international multi-center study, that randomize patients with OHCA of a presumed cardiac or unknown cause to target temperature management at 33°C or normothermia but avoiding fever (37.8°C) for the first 24 hours after the OHCA. The TTM2 study (clinicaltrials.gov Identifier NCT02908308) includes a detailed follow-up of functional outcome, health-related quality of life and neurocognitive function at 6 and 24 months post-arrest. This protocol describes a sub-study within the TTM2 trial that specifically focus on physical activity among the OHCA survivors.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate whether OHCA-survivors have lower levels of self-reported physical activity compared to a non-cardiac arrest (CA) control group who had acute myocardial infarction (MI). Additional aims are to explore potential predictors of physical inactivity (older age, female gender, problems with general physical function, global cognition, mental processing speed/attention, anxiety symptoms, depression symptoms, kinesiophobia, fatigue), and to investigate the relationship between self-reported and objectively measured physical activity among OHCA-survivors.

ELIGIBILITY:
Inclusion Criteria:

* The TTM2 main trial includes adult, unconscious patients with sustained return of spontaneous circulation after cardiac arrest of a presumed cardiac origin. The aim is to include 100-150 OHCA-survivors to the sub-study.

Exclusion Criteria:

* An exclusion criterion for the TTM2 main trial is an unwitnessed cardiac arrest with initial rhythm asystole, temperature at admission <30°C, on extracorporeal membrane oxygenation (ECMO) prior to return of spontaneous circulation (ROSC), obvious or suspected pregnancy, intracranial bleeding and/or severe chronic obstructive pulmonary disease (COPD) on home oxygen.

An additional exclusion criterion for the sub-study is the inability to speak the local language well enough to complete the test without an interpreter. Patients with major cognitive impairment, patients sitting in a wheel chair, Clinical Frailty Score 8 or 9 (very severely frail or terminally ill), active drug abuse and when a face-to face follow-up is not possible will also be excluded.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surviving patients in the TTM2-trial are invited to a structured face-to-face follow-up visit at 180 days (+/- 2 weeks). Survivors at selected sites will be invited to an extended study on physical activity at their follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Physical activity level | 7 months after cardiac arrest
  Questions about physical activity and physical training (patient reported), accelerometer, performance measure

SECONDARY OUTCOMES:
Anxiety and Depression | 7 months after cardiac arrest
  Hospital Anxiety and Depression scale HADS is a self-reported questionnaire with seven questions related to anxiety and seven questions related to depression. Each item on the questionnaire is scored from 0-3. A total sum is calculated for each subscale and the total score range between zero and 21.
Lower extremity strength | 6 months post arrest
  Timed-Stands Test (TST) assess the overall physical function by assessing lower extremity strength
Cognitive impairment | 6 months post arrest
  The Symbol Digit Modalities Test (SDMT) The total amount of correct answers within 90 seconds are calculated. There are normative scores and depending on age and education level
Kinesiophobia | 7 months after cardiac arrest
  Tampa Scale for Kinesiophobia Heart, questionnaire TSK-SV Heart includes17 statements/questions summed into a total score that range from17 to 68. The higher the value, the greater degree of kinsiophobia. Values >37 is considered as a high level of kinesiophobia.
Cognitive impairment | 6 months post arrest
  The Montreal Cognitive Assessment (MoCA). It contains 11 sub-tests of several cognitive domains as executive functioning, short-term memory and delayed recall combined into a total maximum score of 30. A score ≥26 points is considered within the normal range, 25-18 indicate mild impairment, 17-10 indicate moderate impairment, and less than 10 indicate severe cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, MD PhD, Principal Investigator — Lund University; Gisela Lilja, OT PhD, Study Director — Lund University; Tobias Cronberg, PhD MD, Study Director — Lund University; Åsa B Tornberg, RPT PhD, Study Director — Lund University
Locations (8):
- Hans Kirkegaard, Aarhus, Denmark
- Sweden (5):
  - Salgrenska University Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Skane University Hospital Lund, Lund
  - Skane University hospital, Malmo
- United Kingdom (2):
  - Thomas Keeble, Basildon, Essex
  - Mattthew P Wise, Cardiff

REFERENCES:
- [Derived] Heimburg K, Nordstrom EB, Friberg H, Oestergaard LG, Grejs AM, Keeble TR, Kirkegaard H, Mion M, Nielsen N, Rylander C, Segerstrom M, Tornberg AB, Ullen S, Unden J, Wise MP, Cronberg T, Lilja G. Comparison of self-reported physical activity between survivors of out-of-hospital cardiac arrest and patients with myocardial infarction without cardiac arrest: a case-control study. Eur J Cardiovasc Nurs. 2025 Jul 21;24(5):700-709. doi: 10.1093/eurjcn/zvaf032. PMID 39999023
- [Derived] Heimburg K, Lilja G, Tornberg AB, Ullen S, Blennow Nordstrom E, Friberg H, Nielsen N, Ostergaard LG, Grejs AM, Hill H, Keeble TR, Kirkegaard H, Mion M, Rylander C, Segerstrom M, Unden J, Wise MP, Cronberg T. Physical activity after cardiac arrest; protocol of a sub-study in the Targeted Hypothermia versus Targeted Normothermia after Out-of-Hospital Cardiac Arrest trial (TTM2). Resusc Plus. 2021 Jan 29;5:100076. doi: 10.1016/j.resplu.2021.100076. eCollection 2021 Mar. PMID 34223342